CLINICAL TRIAL: NCT00620477
Title: Evaluation of Arthroscopic Reconstruction of the Anterior Cruciate Ligament by One Night Hospital Stay or by Day Surgery: a Randomised, Prospective Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008/068
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Rupture of the Anterior Cruciate Ligament With Instability of the Knee Joint
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): injection in the knee joint with 20 ml of chirocaine 0.125%
  Interventions: Drug: injection in the knee joint with 20 ml of chirocaine 0.125%
- 2 (Placebo Comparator): injection in the knee joint with 20 ml of physiological fluid
  Interventions: Drug: injection in the knee joint with 20 ml of physiological fluid

INTERVENTIONS:
Drug: injection in the knee joint with 20 ml of chirocaine 0.125% — injection in the knee joint with 20 ml of chirocaine 0.125%
  Arms: 1
Drug: injection in the knee joint with 20 ml of physiological fluid — injection in the knee joint with 20 ml of physiological fluid
  Arms: 2

SUMMARY:
Patients who suffered from a rupture of the Anterior Cruciate Ligament with instability of the knee joint, will be treated with an operative ACL-reconstruction. One group of patients will stay one night in the hospital and go home the other day (Group I). The other group of patients will go home the same day of surgery (Group II). All patients will undergo the same arthroscopic reconstruction of the ACL. Anesthesia will be performed on each patient in a classic manner. At the end of the surgery each group of patients will be randomly divided in two subgroups: one group will get an injection in the knee joint with 20 ml of physiological fluid (Group Ia en IIa), the other group will get an injection in the knee joint with 20 ml of chirocaine 0.125%, a widely used pain-medicine (Group Ib and IIb). This will happen in a double blind, randomized way. The whole procedure takes about one hour. After surgery patients are brought to the recovery room and are observed every 30 minutes for the duration of 4 hours. Before being brought to their rooms, patients will have to fill in a VAS: Visual Analogue Scale, to determine their pain. After being brought to their rooms, the patients will have the choice of going home the same day or staying in the hospital for one night, according to the amount of pain they are in. That moment it will be possible to switch groups. Patients who go home the same day of surgery will be contacted by phone the day after to fill in a question form. Patients who were admitted for one night will be seen before their leave to fill in the same question form.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffered from a isolated rupture of the Anterior Cruciate Ligament with instability of the knee joint will be included in the study.
* Patients with a meniscal tear that can be sutured will also be included. Partial meniscectomies are accepted.

Exclusion Criteria:

* Patients with chronic laxity (longer than 9 months), associated collateral laxity (grade III), subtotal or total meniscectomy, infection or inflammatory disease of the knee joint or large cartilage lesion will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07-30 (Actual); Primary Completion 2010-11-03 (Actual); Study Completion 2010-11-03 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | within 4 hours after surgery

SECONDARY OUTCOMES:
Question Form, Visual Analogue Scale | one day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Luc Herregods, MD, PhD, Principal Investigator — University Hospital, Ghent; Fredrik Almqvist, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be